CLINICAL TRIAL: NCT01228942
Title: A Prospective Trial of COXEN Chemotherapy Prediction in Persistent and Recurrent Ovarian, Fallopian Tube, and Peritoneal Carcinomas
Brief Title: A Prospective Trial of COXEN Chemotherapy Prediction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding/resources
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Linda R Duska, Medical Attending, University of Virginia
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 15248
Record Dates: First submitted 2010-10-20; First posted 2010-10-27 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms
Keywords: ovarian cancer; fallopian tube cancer; primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platinum Sensitive (Other): Treatment with platinum-based therapy; COXEN prediction model chooses secondary agent if doublet
  Interventions: Device: COXEN analysis for chemotherapy prediction
- Platinum resistent (Other): single agent based on Coxen prediction model
  Interventions: Device: COXEN analysis for chemotherapy prediction

INTERVENTIONS:
Device: COXEN analysis for chemotherapy prediction — Using the affymetrix genechip along with the COXEN algorithm the subject's treatment will be determined
  Other Names: Affymetrix genechip

SUMMARY:
The purpose of this study is to determine if the COXEN algorithm, using the diagnostic device Affymetrix GeneChip, is able to predict which chemotherapies will be best for treatment of recurrent or persistent ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
The current proposal seeks to apply and extend this novel genomic prediction technique to finding better chemotherapeutic options for recurrent ovarian cancer using individual patients' gene-expression signatures of chemosensitivity. The utility of the COXEN technique has been validated and found to accurately predict 1) the chemosensitivity of an independent panel of 40 bladder cancer cell lines; 2) activity of each of the >45K candidate compounds in the NCI-60 drug screening database, which resulted in the identification of a highly-effective novel compound for bladder cancer and patients' responses and survival on 12 historical clinical trials of combination chemotherapy. In particular, the GEMs of breast cancer can be used to stratify both clinical response and overall patient survival with a striking difference between the predicted responders vs. predicted non-responders in 5 independent chemotherapeutic trials of breast cancer. The next step is to test the prediction model in recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18
* diagnosis of recurrent, persistent, refractory ovarian, fallopian or primary peritoneal cancer
* tumor tissue, ascites or pleural fluid available for biopsy
* life expectancy greater than 6 months

Exclusion Criteria:

* patients with borderline or low malignant histologies
* patients with a history of other malignancies within last 5 years

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
overall response rate | 12 months
  patient will have CT scans and CA 125 drawn to track response to chemotherapy

SECONDARY OUTCOMES:
overall survival | subject lifetime
  patient will be tracked for life

CONTACTS AND LOCATIONS:
Overall Officials: Linda Duska, MD, Principal Investigator — University of Virginia